CLINICAL TRIAL: NCT02567630
Title: Early Childhood Constraint Therapy for Sensory/Motor Impairment in Cerebral Palsy
Brief Title: Early Childhood Constraint Therapy in Cerebral Palsy
Acronym: APPLES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Nathalie Maitre, Director NICU follow up program, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB15-00547
Record Dates: First submitted 2015-08-26; First posted 2015-10-05 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Soft Mitt Constraint Therapy for Sensory/Motor Impairment in Cerebral Palsy — The CIMT intervention includes 3 components: (1) placement of a removable soft constraint for ½ each day, with a non-invasive wear monitor (2) demonstration and prescribed home-use of a sensory kit (3) and a reach/grasp tool. The intervention lasts 4 weeks as has been published in older children as well as used in infant trial descriptions.

SUMMARY:
This is a prospective interventional study involving young children who will all receive non-invasive, passive assessments of sensory and motor function. In addition a subpopulation of young children with cerebral palsy will participate in a randomized controlled trial of constraint-induced movement therapy, a routinely prescribed therapy used in clinical practice for children with motor difficulties. The study attempts to apply a rigorous scientific approach to study a widely used but poorly studied practice. The design is an RCT with wait-list controls to allow all children to benefit from the therapy, even if they are randomized to the control group. All children, regardless of group allocation will continue with their standard of care occupational and physical therapy throughout the study.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability in childhood.1 It affects 3.6/100 children in the US2 with ~10,000 new diagnoses every year. The prevalence of CP in developing countries is estimated to be ~5-10 times greater. CP is a disorder resulting from sensory and motor impairments due to perinatal brain injury, with lifetime consequences that range from poor adaptive and social function to communication and emotional disturbances,9 all contributing to a shortened life expectancy. The societal costs are difficult to estimate but the financial burden is well over $1 M per life affected. A growing number of evidence-based therapies aim to improve gross motor function through changes in body structures and function in children with CP (e.g. hip surveillance, surgery). However, infants with CP have a fundamental disadvantage in recovering motor function: they do not receive accurate sensory feedback from their movements, leading to neglect of an affected extremity and difficulty learning new movements, a process called developmental disregard (DD). As a consequence, even children who receive time- and resource-intensive standard therapies have stable or declining motor function and developmental trajectories that do not "catch up" to those of typically developing children. DD can then lead to school-age learning problems, decreased participation in physical and social activities and costly long-term mental and physical morbidities.

Constraint-Induced Movement Therapy (CIMT) is one of the few effective neurorehabilitative strategies shown to improve upper extremity motor function in adults and older children with CP, potentially overcoming developmental disregard. It is mainly applicable to CP patients who are diagnosed with asymmetric or hemiparetic forms of the disorder, in which one side of the body is more affected than the other. CIMT is based on the premise that preferential use of an affected upper extremity (by constraining the less affected one), and shaping with repetition of movement by skilled therapists, can overcome neglect and restore function of that extremity.

The investigators are conducting a randomized trial of CIMT in children with CP using a wait-list control group. This design allows every child with CP to eventually receive the treatment and avoids issues of equipoise. The RCT portion of the study extends only for a 7-month period, from baseline to 6 months after the 1-month CIMT ends. For CP wait-listed controls, the study continues for 6 months following the CMIT intervention, separate from the completed RCT. We will reference data from both groups to a cohort of typically developing (TD) children to determine developmental trajectories.

ELIGIBILITY:
Inclusion Criteria:

* CP children (n=72): Inclusion criteria will be diagnosis of hemiparetic or asymmetric CP as determined by published algorithms and neurologic exam.
* TD children (n=144): Inclusion criteria will be GA and sex-matched compared to the CP group, with CA at assessment matched to the CP group at baseline (72 children) and at the 7-month assessment (72 children). Exclusion criteria will be any motor or sensory impairment as defined by neurologic exam and/or scaled motor scores below 8 for CA on the Bayley III and cognitive impairment or delays as described for the CP group.

Exclusion Criteria:

* CP children: exclusion criteria will be CP with Gross Motor Function Classification Score (GMFCS) of 4-5, corresponding to poor or absent mobility and neck control; receipt of Botox to the affected extremity within 3 months of study entry; or scores of <70 on the Bayley Scales of Infant Development (Bayley III) cognitive composite.
* TD children: Exclusion criteria will be any motor or sensory impairment as defined by neurologic exam and/or scaled motor scores below 8 for CA on the Bayley III and cognitive impairment or delays as described for the CP group.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Estimated)
Dates: Start 2015-10-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Kinematics of reach | Change from Baseline to Post intervention (1 month), and 6 months later
  We will use a motion analysis system tracks reflective markers at a rate of 240 Hz with spatial precision at the 1-mm level to capture movement in three-dimensional space. Markers will be positioned bilaterally on the head of the second metacarpal bone and on the object. Tracker software will be used to determine the three-dimensional position of the hand as it approaches each object, and to construct segments, angles and moments using Matlab software.
  For each trial, approach velocity and movement units (marked by changes in speed or position) will be calculated. A single movement unit is defined as the portion of reach between one acceleration and another. The sum composite of movement units in one reach attempt is defined as smoothness. The motion tracking data will also be used to determine the time from presentation to first contact, time from first contact to grasp and approach velocity on the unilateral task.
Somatosensory processing measurement by ERP | Change from Baseline to Post intervention (1 month), and 6 months later
  A high-density array of 128 electrodes embedded in soft sponges (Geodesic Sensor Net, EGI, Inc., Eugene, OR) will be used to record ERPs with a sampling rate of 1000 Hz, filters set to 0.1-400 Hz. All electrodes will be referred to Cz and re-referenced offline to an average reference. Recording of brainwaves will be controlled by Net Station (v. 4.3; EGI, Inc., Eugene, OR). E-Prime (v. 2.0, PST, Inc., Pittsburgh, PA) software will control stimulus delivery. Air puffs will be delivered using a custom-made apparatus with two flexible nozzles, one positioned approximately 0.5" below the palm of hand secured in a molded soft holder (puff condition), the other placed in proximity but directed away (sham condition). The pressure at the skin surface is 5 psi, or less than the pressure of the smallest microfilament used to test for neuropathies. For each hand, 60 puffs will be presented randomly interspersed with 60 sham trials.
Bayley Scales of Infant and Toddler Development (Bayley III) - 3rd Edition | Change from Baseline to Post intervention (1 month), and 6 months later
  The Bayley III is the gold standard for the evaluation of former NICU graduates, and we have extensive experience using it in the Follow-Up Clinic. The motor scales provide a developmental and functional assessment, address unimanual as well as bimanual skills, are normed against a large population and designed to be adjusted for varying degrees of prematurity.
  The Bayley fine motor items for 6-24 months (score range: 0-42) measure prehension, motor planning, grasping patterns, and eye-hand coordination. The examiner is masked to intervention vs. control group membership and administers the fine motor subscale twice, repeating unilateral items for right and left hands. Most (about 80%) of the Bayley fine motor items for infants aged 6 to 24 months require unilateral reach and grasp.
  In addition to standard testing, separate scores will be obtained to characterize the difference between more and less affected extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie L Maitre, MD, PhD, Principal Investigator — Nationwide Childrens hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Maitre NL, Jeanvoine A, Yoder PJ, Key AP, Slaughter JC, Carey H, Needham A, Murray MM, Heathcock J; BBOP group. Kinematic and Somatosensory Gains in Infants with Cerebral Palsy After a Multi-Component Upper-Extremity Intervention: A Randomized Controlled Trial. Brain Topogr. 2020 Nov;33(6):751-766. doi: 10.1007/s10548-020-00790-5. Epub 2020 Aug 3. PMID 32748303
- [Derived] Chorna O, Heathcock J, Key A, Noritz G, Carey H, Hamm E, Nelin MA, Murray M, Needham A, Slaughter JC, Maitre NL. Early childhood constraint therapy for sensory/motor impairment in cerebral palsy: a randomised clinical trial protocol. BMJ Open. 2015 Dec 7;5(12):e010212. doi: 10.1136/bmjopen-2015-010212. PMID 26644127